CLINICAL TRIAL: NCT03617614
Title: Evaluation of the Medical Psychiatry Alliance Senior's Outpatient Collaborative Care Project
Acronym: MPASOP
Status: Completed | Type: Observational
Sponsor: Trillium Health Centre (Other)
Collaborators: Centre for Addiction and Mental Health (Other); Medical Psychiatry Alliance (Other)
Responsible Party: Principal Investigator, Judith Versloot, Research Lead (PhD), Trillium Health Centre
Other Study IDs: TrilliumHC
Record Dates: First submitted 2018-07-19; First posted 2018-08-06 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — engage 8200

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Collaborative Care Model: Participants who received care from the Medical Psychiatry Alliance Seniors Outpatient Collaborative Care Program at Trillium Health Partners.
  Interventions: Behavioral: Collaborative Care Model
- Mood Consult: Participants who received a one time mood consultation at the Centre for Addiction and Mental Health.
  Interventions: Behavioral: Mood Consultation

INTERVENTIONS:
Behavioral: Collaborative Care Model — Trained care managers (CM) work collaboratively with patients, caregivers, and primary care providers to provide education, care navigation and behavioral activation. The latter includes a stepped psychotherapy intervention called ENGAGE, that focuses on "reward exposure" engagement in meaningful, rewarding activities for patients. Patients (home) visits are delivered over a period of 6 to 16 weeks. Progress is assessed with standardized measures for depression (PHQ-9), anxiety (GAD-7) and functioning (WHO-DAS). Furthermore, patients are presented by the CM at Systematic Case Review meetings where an integrated team of medical, psychiatric and allied health professionals work collaboratively to review the patient's goals and treatment to formulate a care plan and recommendations.
  Other Names: ENGAGE
  Groups: Collaborative Care Model
Behavioral: Mood Consultation — A meeting with a psychiatrist to do assessment, provide education and make recommendations regarding the care of the patient for the Primary Care Provider.
  Groups: Mood Consult

SUMMARY:
This study evaluates the effectiveness of a collaborative care model designed to treat frail seniors with both a mental (anxiety and/or depression) and a physical health condition impacting function with a comparison group that receives a psychiatric mood consult and a letter of recommendation but who are mainly cared for by their PCP.

DETAILED DESCRIPTION:
Literature suggests seniors with co-existing mental and physical health concerns encounter challenges with accessing care including limited availability of geriatric specialists, inadequate navigational support, disjointed communication, and limited provider knowledge/ capacity to manage these complex patients. In conjunction with primary care, a new program was created to assist in addressing these concerns. A novel collaborative care model was developed integrating Geriatric Medicine and Geriatric Psychiatry anchored in primary care, where primary care remains the most responsible provider. Care managers (CMs) work with seniors in the community, for up to 16 weeks, who have at least one chronic health condition affecting function and depressed mood and/or anxiety. The care model focusses on 4 main components: integrated therapeutic care management, systematic case reviews (SCRs), integrated care planning, and education/capacity building. CMs provide comprehensive assessments, system navigation, monitoring using symptom rating scales, and a problem solving psychotherapy for seniors using reward exposure to form action plans (ENGAGE). CMs present cases weekly at SCRs, where the team includes a geriatrician, geriatric psychiatrist, primary care, and allied health. Recommendations are made then sent to the PCP for implementation. In the current evaluation study we will compare levels of depression, anxiety and functioning of seniors receiving the collaborative care model with those receiving a one time mood consultation.

ELIGIBILITY:
Inclusion Criteria:

* Depressive mood PHQ-9 >9 or anxiety GAD-7 >9
* One or more chronic medical condition(s) impacting function
* Had a one time mood consultation at CAMH or has been a patient in the Medical Psychiatry Alliance Senior Outpatient Program
* Able to speak English

Exclusion Criteria:

* Moderate to severe cognitive decline
* Positive psychotic symptoms
* Active suicidal ideation or attempt within the last year
* Psychiatric admission within the last year

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Seniors discharged from the Medical Psychiatry Alliance Senior Outpatient Program or Seniors that received a one time mood consultation at CAMH
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9) from baseline to 12 months after discharge | Baseline to 12 months after discharge
  The Patient Health Questionnaire (PHQ-9) is a 9-item questionnaire that is used for screening, diagnosing, monitoring, and measuring the severity of depression. Each item can be answered on a 4 point scale running from 0= 'not at all' to 3= 'nearly every day'. The total score ranges from 0-27 where 0 is no depression and 27 is severe depression.

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder 7-item (GAD-7) from baseline to 12 months | Baseline to 12 months after discharge
  The Generalized Anxiety Disorder 7-item (GAD-7) is a 7-item questionnaire that is used for screening, diagnosing, monitoring, and measuring the severity of anxiety. Each item can be answered on a 4 point scale running from 0= 'not at all sure' to 3= 'nearly every day'. The total score ranges from 0-21 where 0 is no anxiety and 27 is severe anxiety.
Change in World Health Organization Disability Assessment Schedule 2.0 (WHODAS) from baseline to 12 months | Baseline to 12 months after discharge
  The WHODAS is a practical generic assessment instrument that is used to measure health and disability. The WHODAS captures level of functioning in six domains: cognition, mobility, self-care, getting along and life activities. The 12-item questionnaire version asks about difficulties due to patient health conditions. Patients answer 12 questions within the 6 domains and select the best option of 5 answer categories: 1=none, 2=mild, 3=moderate, 4=severe, 5=extreme or cannot do. The total sum of the questions range between 12-60. and is than divided by 12 to determine where the patient falls on "none to extreme or cannot do" (range 1-5) scale .
Patient satisfaction with care | 12 months after discharge
  The question that will be asked is: 1) I think the services provided at CAMH/THP were of high quality. The answer category is a 5-point likert rating scale running form 5=strongly agree to 0=strongly disagree. Score range 0= not at all satisfied to 5= very satisfied.
Healthcare Utilization in the previous 3 months | 12 months after discharge
  The participants will be asked 6 questions about if the participant has seen a family physician, social worker, psychiatrist, psychologist and/or visited the emergency department and/or has been admitted to the hospital in the past 3 months. The number of health care providers seen will be summed to a total score that ranges from 0-6 where 0 represents no health care utilization and 6 represent high healthcare utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Versloot, PhD, Principal Investigator — Trillium Health Partners
Locations (2):
- Canada (2):
  - Trillium Health Partners, Mississauga, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.